CLINICAL TRIAL: NCT03326466
Title: The Subacromial Shoulder Pain and Central Nervous System Sensitization Trial (SAP-CNSS):Central Nervous System Sensitization, Muscle Function, and Pain Profiling in Patients With Subacromial Pain and in Healthy Controls.
Brief Title: Muscle Function, Central Nervous System Sensitization, and Pain Profiling in Patients With Subacromial Pain (SAP-CNSS).
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Physical Medicine and Rehabilitation Research - Copenhagen (PMR-C). (Unknown); Metropolitan University College (Other); Center for Neuroplasticity and Pain (CNAP). (Unknown); National Research Center for the Working Environment. (Unknown)
Responsible Party: Principal Investigator, Bjarki Haraldsson, MSc, PhD, Hvidovre University Hospital
Other Study IDs: SAP-CNSS
Record Dates: First submitted 2017-10-12; First posted 2017-10-31 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Subacromial Impingement Syndrome; Central Nervous System Sensitization
Keywords: Subacromial Impingement Syndrome; Central Nervous System Sensitization; Muscle Function; EMG; Force Steadiness; CUFF Algometry; Manual Algometry; Pain; Maximal Voluntary Isometric Contraction
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with SAP
- Healthy Controls

SUMMARY:
In this case-control study, the investigators compare shoulder muscle function, pain, and central nervous system sensitization in patients with Subacromial Pain (SAP) to that in healthy controls. The investigators also examine if a relationship exists between shoulder symptom duration and central sensitization, shoulder muscle function and shoulder pain distribution in patients with SAP.

DETAILED DESCRIPTION:
Subacromial pain (SAP), also referred to as subacromial impingement syndrome, is characterized by pain in the shoulder joint, which is aggravated by elevation of the arm and / or during overhead activities. Subacromial pain has been suggested to be an "end station" to numerous pathologies of the shoulder and can be considered to include a variety of symptoms, and not to be seen only as a single diagnosis. In Denmark, SAP is frequently reported as a cause of pain in the shoulder joint, and based on studies from Sweden and the Netherlands, is estimated to cost the Danish society around 1.35 billion. DKK annually.

The primary aim of this study is to compare central nervous system sensitization (central sensitization), shoulder muscle function and shoulder pain distribution in patients with subacromial pain to that in pain free healthy matched controls.

The secondary aim of this study is to investigate if (symptom) dose/response relationships exist between shoulder symptom duration and: central sensitization, shoulder muscle function and shoulder pain distribution in patients with subacromial pain.

Although the present study is exploratory, it is the working hypothesis that i) patients with subacromial pain have increased central sensitization, reduced shoulder muscle function, and increased pain distribution when compared to healthy controls, and ii) symptom dose/response relationships exist, indicated by increased central sensitization, reduced shoulder muscle function, and increased pain distribution with longer symptom duration in patients with subacromial pain.

The methodology includes: surface EMG recordings to quantify shoulder muscle activity; dynamometry to quantify maximal voluntary contraction force and submaximal isometric force steadiness; mechanical and computer-controlled algometry to quantify CNS sensitization; computerized pain drawings to quantify pain distribution; and patient-reported assessments of shoulder pain (SPADI) and catastrophizing (PCS).

The study does not include any intervention.

The present study is considered exploratory and the first in a line of studies using these outcome measures in this patient population. All outcomes listed below are valued equally, as the study is exploratory. All analyses will be used to indicate effect sizes in order to plan for subsequent follow-up studies.

Although the study is considered exploratory, the statistical approach includes the pre-defined primary and secondary analyses outlined below.

Primary analysis: The primary analysis will compare 36 included patients to 36 matched healthy controls regarding the 3 main outcomes: shoulder muscle function, CNS sensitization and shoulder pain distribution.

Secondary analysis: The secondary analysis will compare the three subgroups of patients differing in their symptom duration (0.5-3 months of pain, 3-6 months of pain and +6 months of pain), regarding the 3 main outcomes: CNS sensitization, shoulder muscle function, and shoulder pain distribution, to indicate (symptom) dose/response relationships, using descriptive statistics. The symptom duration groups may be redefined, if recruitment is slow for one or more of the groups outlined above.

Collaborators:

Thomas Bandholm, PT, Professor, PhD. PMR-C.

Kristian Thorborg, PT, Associate Professor, PhD. Department of Clinical Medicine, University of Copenhagen, Amager/Hvidovre Hospital.

Thomas Graven-Nielsen, Professor, Director. CNAP.

Michael Skovdal Rathleff, PT, PhD. Department of Health Science and Technology Aalborg University.

Shellie Boudreau, Associate Professor. Department of Health Science and Technology Aalborg University.

Louisa Wilquin, PT. School of Physiotherapy, Metropolitan University College Copenhagen.

Mikkel Bek Clausen, PT, PhD-fellow. Department of Clinical Medicine, University of Copenhagen, Amager/Hvidovre Hospital.

Markus Due Jacobsen, PhD. National Research Center for the Working Environment.

Lars Andersen, Professor, PhD. National Research Center for the Working Environment.

ELIGIBILITY:
Inclusion Criteria:

* Have had SAP during the last two weeks or more.
* Have positive results from minimum 3 out of 5 clinical tests.
* Have experienced pain ranking 4 or above on the VRS scale within the last 7 days.
* Are able to speak and understand Danish.
* Have given informed consent to participate in the study after they have fully understood the content of the study.

Exclusion Criteria:

* Have acquired traumatic shoulder injury, and this is onset/cause for current shoulder pain, e.g. fall on shoulder.
* Have received a corticosteroid injection within the last six weeks.
* Report having had a shoulder fracture within 6 months.
* Report having had surgery on the affected shoulder.
* Report having radiologically verified glenohumeral osteoarthritis.
* Have a luxation or sub-luxation of the glenohumeral or the acromioclavicular joint, clinically suspected labrum lesion, clinically suspected complete traumatic tear of the rotator cuff, frozen shoulder, suspected competing diagnoses (i.e. rheumatoid arthritis, cancer, neurological disorders, and fibromyalgia).
* Have a history of diagnosed major psychiatric disorder.
* Have a history of illicit drug use; be currently abusing alcohol or currently withdrawing from alcohol abuse.
* Have a history of heart disease.
* Are pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subacromial Pain.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximal Voluntary Strength. | Baseline assessment, no follow-up (cross-sectional study).
  Unit of Measure: Nm/Kg.
Submaximal Voluntary Force Steadiness | Baseline assessment, no follow-up (cross-sectional study).
  Unit of Measure: Nm/Kg.
Maximal EMG | Baseline assessment, no follow-up (cross-sectional study).
  Unit of Measure: mV/s. Will be recorded during the measurement of Maximal Voluntary Strength.
Submaximal EMG. | Baseline assessment, no follow-up (cross-sectional study).
  Unit of Measure: mV/s. Will be recorded during the Measurement of Force Steadiness.
Central Nervous System Sensitization - Manual Algometry. | Baseline assessment, no follow-up (cross-sectional study).
  Unit of Measure: kPa/s
Central Nervous System Sensitization - Cuff Algometry. | Baseline assessment, no follow-up (cross-sectional study).
  Unit of Measure: kPa/s.
Patient Reported Outcome - Pain Mapping. | Baseline assessment, no follow-up (cross-sectional study).
  Subject will draw their pain as accurately as possible on a high resolution 3D body schema.
  Area of Pain is quantified as total number of pixels, and will be expressed as percentage of body area.
Patient Reported Outcome - Shoulder Pain And Disability Index (SPADI). | Baseline assessment, no follow-up (cross-sectional study).
  Questionnaire contains 13 items with a possible score from 0-100 (0=no disability).
Patient Reported Outcome - Pain Catastrophizing Scale (PCS). | Baseline assessment, no follow-up (cross-sectional study).
  Questionnaire contains 13 items with a possible score 0-52. Higher score indicates higher level of pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bandholm, PhD, Study Chair — Professor, Head of Research, PMR-C.
Locations (1):
- Hvidovre University Hospital, Hvidovre, Sealand, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We intend to make the data set - containing de-identified individual-patient data - publically available no later than 6 months after publication, consistent with the recent proposal from the International Committee of Medical Journal Editors (ICMJE), if it complies with national regulations, e.g. the Danish Data Protection Agency.